CLINICAL TRIAL: NCT07194564
Title: Acute Effect Assessment of a Self-corrective Exercise on Electromyography and Spine Deviation in Adolescent Idiopathic Scoliosis
Brief Title: Acute Training Effect Assessment in Adolescent Idiopathic Scoliosis
Acronym: AcuteEMGAIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yifan HUANG, Postdoctoral Fellow, The University of Hong Kong
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UW24-747
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Adolescence Idiopathic Scoliosis; AIS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Exercise (Active Comparator): Participants perform a standard exercise that does not include self-correction elements. This serves as the control condition for comparison.
  Interventions: Behavioral: Control Exercise
- Self-corrective Exercise (Experimental): Participants perform a self-corrective exercise designed to improve spinal alignment and muscle activity.
  Interventions: Behavioral: Self-corrective Exercise

INTERVENTIONS:
Behavioral: Control Exercise — A standard exercise without self-correction, performed by all participants as the control condition.
  Arms: Control Exercise
Behavioral: Self-corrective Exercise — A self-corrective exercise intervention targeting improved postural alignment and muscle activation.
  Arms: Self-corrective Exercise

SUMMARY:
This study aims to assess the immediate effects of a self-corrective exercise on muscle activity and spinal alignment in adolescents with idiopathic scoliosis. Eligible participants will undergo clinical assessments of spine deviation and surface electromyography (EMG) before and after a single session of guided self-controled and self-corrective exercise. The findings may help inform rehabilitation strategies for adolescent idiopathic scoliosis.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) involves three-dimensional spinal deformity and asymmetric paraspinal muscle activation. Scoliosis-specific, self-corrective exercises are widely used in conservative care, but their immediate neuromuscular and postural effects after a single guided session remain insufficiently characterized.

This prospective pre-post study will enroll adolescents with radiographically confirmed AIS for one clinic visit. After eligibility confirmation and consent/assent, participants will complete baseline assessments, perform a standardized, therapist-guided self-controlled, self-corrective exercise tailored to curve pattern, and then repeat the same assessments immediately afterward. The protocol emphasizes axial elongation, active self-correction delivered within a brief supervised session.

The primary purpose is to quantify immediate changes in spinal alignment and paraspinal muscle activity to explore potential mechanisms of action and inform refinement of rehabilitation strategies for AIS. Feasibility and tolerability will be monitored during the single visit. No additional imaging is required beyond existing clinical records. Findings will be disseminated through scientific channels to guide future conservative management and hypothesis generation for subsequent controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* adolescent males and females with AIS
* being aged 11 to 19 years

Exclusion Criteria:

* having a nonidopathic etiology of scoliosis
* history of spinal surgery; spine trauma (e.g., fracture or motor vehicle accident)
* metal implants (e.g., pacemaker)
* not capable of understanding and completing our motor tasks
* experiencing severe dermatological conditions or have open wounds at electrode placement sites.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-08-03 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Back muscle symmetry assessed by surface electromyography (sEMG) using the Asymmetry Index (ASI). | Immediately after each exercise session.
  Surface EMG signals will be recorded from bilateral back muscles to assess muscle symmetry. The the Asymmetry Index (ASI) ranges from 0 to 1, where 1 indicates complete asymmetry and 0 indicates perfect symmetry. Higher values indicate greater asymmetry.

SECONDARY OUTCOMES:
Vertical line deviation (VLD) of spinous processes and sacrum in the coronal plane (posterior view) | Immediately after each exercise session
  The deviation of spinous processes and sacrum from the vertical line will be measured in the coronal plane from a posterior view.

CONTACTS AND LOCATIONS:
Locations (1):
- the Duchess of Kent Children's Hospital; the University of Hong Kong', Hong Kong, Remote, Hong Kong

IPD SHARING:
Plan to Share IPD: No